CLINICAL TRIAL: NCT03793946
Title: A Digital Antimicrobial Stewardship Smartphone Application to Combat AMR: the AB-assistant: an International, Multicenter Stepped-wedge Cluster Randomized Trial
Brief Title: A Digital Antimicrobial Stewardship Smartphone Application to Combat AMR: the AB-assistant
Acronym: AB-assistant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Annelies Verbon (Other)
Collaborators: Erasmus Medical Center (Other); University Hospital, Geneva (Other); Uppsala University Hospital (Other); University of Calgary Cumming School of Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Annelies Verbon, Prof. dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZonMw_549003001
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Anti-Infective Agents; Mobile Applications; Quality Improvement; Antimicrobial Stewardship
Keywords: Drug Resistance, Microbial; Multicenter Study; Decision Support Systems, Clinical

STUDY DESIGN:
Intervention Model Description: International, multicenter stepped-wedge cluster randomized trial
Who Masked: Outcomes Assessor
Masking Description: Masking of care providers and investigators is not feasible. Outcome assessors and data analysts will be blinded to the study arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB-assistant (Experimental): Use of the AB-assistant app by physicians in intervention wards.
  Interventions: Other: AB-assistant
- Standard antimicrobial stewardship (No Intervention): Physicians on these wards will use conventional ways to assess local guidelines to prescribe antimicrobials.

INTERVENTIONS:
Other: AB-assistant — The AB-assistant is an antimicrobial stewardship smartphone application that offers local antimicrobial guidelines to physicians currently assessed per website or paper/digital booklet.
  Arms: AB-assistant

SUMMARY:
Optimal prescribing of antimicrobials is becoming increasingly challenging because of the growing complexity of guidelines and constantly changing distribution of infectious pathogens. Prescribing antimicrobials appropriately according to local guidelines optimizes therapy for the individual patient and reduces the emergence of resistance. By adapting and evaluating a smartphone based app containing local guidelines we aim to study appropriate prescribing of antimicrobials by physicians in three hospitals (Netherlands, Sweden and Switzerland).

DETAILED DESCRIPTION:
Rationale: Antimicrobials are an indispensable part of modern medicine. However, optimal prescription of these agents is becoming increasingly challenging because of the growing complexity of guidelines, and constantly changing epidemiology of infectious pathogens. Moreover, due to local variations in the prevalence of certain pathogens and antimicrobial resistance (AMR), antimicrobial choices need to be tailored to local epidemiology. Improvement of antimicrobial use, in particular prevention of overuse and suboptimal use of antimicrobials, through antimicrobial stewardship (AMS) programs is increasingly regarded as indispensable, both to optimize therapy for the individual patients as well as to reduce emergence and spread of AMR. With the widespread use of electronic health records (EHR) and handheld electronic devices in hospitals, informatics-based AMS interventions hold great promise as tools to improve antimicrobial prescribing. However, they are still underdeveloped, understudied and underutilized.

Objective: The study aims to adapt and evaluate the "AB-assistant", a smartphone based digital stewardship application that is customizable to local guidelines by local antibiotic stewards and therefore has the potential to be used worldwide, including in low- and middle-income countries.

Study design: The existing North American Spectrum app (SpectrumMD; Canada) will be adjusted and translated for the European market. During a usability study physicians will use the app for two weeks followed by individual interviews to determine facilitators and barriers of app use. Based on the results of these interviews the app will be adjusted if necessary. After adaptation and usability testing, thereafter the AB-assistant app will be evaluated in an international, multicentre, randomized clinical trial involving centres in 3 countries in different settings with appropriate antimicrobial use as a primary outcome. In a stepped wedge cluster randomized trial, wards will be randomised after stratification for specialty. At baseline a 2-week measurement period will be done, followed by the introduction of the intervention to 6 wards (in 3 hospitals) with a 4-week interval with 6 inclusion periods. This cycle will be repeated with the inclusion of all new intervention wards. We include the 36 wards in total during the 6 inclusion phases and at the end of the inclusion time we allow use of the app by everyone, also wards not included in the study.

ELIGIBILITY:
Inclusion Criteria:

Cluster level (wards):

• Medical and surgical wards.

Physician level:

• All physicians involved in antibiotic prescribing decisions in the participating wards.

Patient level:

• All patients hospitalized in the participating wards >= 18 years of age to whom systemic antimicrobials are prescribed.

Exclusion Criteria:

Cluster level (wards):

* Outpatient clinics
* Psychiatry wards
* ICU

Physician level:

• None

Patient level:

• None

Treatment level:

• Surgical and medical prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Appropriate empirical antimicrobial therapy | 12 months
  According to predefined criteria

SECONDARY OUTCOMES:
Total prescription of antimicrobial drugs | 12 months
  In defined daily dose (DDD)/admission
Total prescription of antimicrobial drugs per AWaRe category in DDD/admission | 12 months
  Per AWaRe category in DDD/admission
Antimicrobial costs | 12 months
  Total costs of antimicrobial drugs administered
Length of hospital stay (LOS) | 12 months
  (LOS)
In-hospital mortality | 12 months
  All cause in-hospital mortality
Hospital readmission within 30 days of discharge | 12 months
  Unplanned hospital readmissions within 30 days after discharge
Transfer to intermediate care or ICU | 12 months
  % of admissions transferred to intermediate care or ICU after initial non-intermediate care or non-ICU admission
Incidence Clostridium difficile infections (CDI) | 12 months
  Incidence of healthcare facility onset Clostridium difficile
Incident clinical cultures with multi-drug resistant organisms (MDRO) | 12 months
  Incidence of clinical cultures with multidrug resistant organisms (methicillin-resistant Staphylococcus aureus (MRSA), Extended spectrum beta-lactamase producing Enterobacteriaceae (ESBL-E), carbapenemase-producing Enterobacteriaceae (CPE), vancomycin-resistant enterococci (VRE), multidrug resistant P. aeruginosa) denominated per 1000 patient days and admissions
Uptake of the AB-assistant | 12 months
  Total users and number of sessions per user, time spent per session, time spent per screen, number of times each screen is viewed.
Actual use of AB-assistant and experiences while using it | 12 months
  Questionnaire
Number of infectious diseases consultations | 12 months
  Total amount of infectious diseases consultations

CONTACTS AND LOCATIONS:
Overall Officials: B D Huttner, MD, MS, Principal Investigator — University Hospital, Geneva; T Tängdén, MD, PhD, Principal Investigator — Uppsala University; John Conly, Prof. Dr., Principal Investigator — University of Calgary Cumming School of Medicine
Locations (4):
- University of Calgary Cumming School of Medicine and Alberta Health Services, Department of Medicine, Calgary, Alberta, Canada
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- Uppsala University, Dept of Medical Sciences, Uppsala, Sweden
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data will be made publicly on request available from the time of publication or within a reasonable time period of the experiments being completed. General project data and metadata will be included in the supplementary data of published articles if needed and or shared through university repositories.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Helou RI, Catho G, Faxen L, Hulscher M, Teerenstra S, Conly J, Huttner BD, Tangden T, Verbon A. Impact of a smartphone application for appropriate antibiotic prescribing at three tertiary hospitals: an international, multicentre stepped-wedge cluster randomized trial. Clin Microbiol Infect. 2025 Jul;31(7):1172-1179. doi: 10.1016/j.cmi.2025.02.026. Epub 2025 Mar 1. PMID 40032084
- [Derived] Helou RI, Catho G, Peyravi Latif A, Mouton J, Hulscher M, Teerenstra S, Conly J, Huttner BD, Tangden T, Verbon A. Study protocol for an international, multicentre stepped-wedge cluster randomised trial to evaluate the impact of a digital antimicrobial stewardship smartphone application. BMJ Open. 2020 Jun 4;10(6):e033640. doi: 10.1136/bmjopen-2019-033640. PMID 32503867